CLINICAL TRIAL: NCT00079027
Title: A Randomized Clinical Trial Evaluating the Benefits of Doxorubicin Chemoembolization Versus Systemic Doxorubicin in Patients With Unresectable, Advanced Hepatocellular Carcinoma
Brief Title: Doxorubicin By Infusion or Chemoembolization in Treating Patients With Advanced Unresectable Hepatocellular Carcinoma (Liver Cancer)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital Birmingham (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000353298; CRUK-HEP-1; EU-20340; ISRCTN78345798
Record Dates: First submitted 2004-03-08; First posted 2004-03-09 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2007-05

CONDITIONS: Liver Cancer
Keywords: advanced adult primary liver cancer; adult primary hepatocellular carcinoma
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Doxorubicin

INTERVENTIONS:
Drug: doxorubicin hydrochloride
Procedure: hepatic artery embolization

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as doxorubicin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping the cells from dividing. Chemoembolization kills tumor cells by blocking the blood flow to the tumor and keeping chemotherapy drugs near the tumor. It is not yet known whether doxorubicin is more effective with or without chemoembolization in treating unresectable hepatocellular carcinoma (liver cancer).

PURPOSE: This randomized phase III trial is studying doxorubicin given by infusion to see how well it works compared to doxorubicin given by chemoembolization in treating patients with advanced liver cancer than cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the survival of patients with advanced unresectable primary hepatocellular carcinoma treated with intravenous doxorubicin hydrochloride vs doxorubicin hydrochloride chemoembolization.

Secondary

* Compare the response rate in patients treated with these regimens.
* Compare time to progression in patients treated with these regimens.
* Compare the toxicity of these regimens in these patients.
* Compare the quality of life of patients treated with these regimens.
* Compare the health economic implications of these regimens in these patients.

OUTLINE: This is a randomized, controlled, multicenter study. Patients are stratified according to participating center, stage of disease, and alpha-fetoprotein levels (< 500 ng/mL vs ≥ 500 ng/mL). Patients are randomized to 1 of 2 treatment arms.

* Arm I (control arm): Patients receive doxorubicin hydrochloride IV over 3-5 minutes on day 1. Treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.
* Arm II (chemoembolization arm): Patients undergo transarterial chemoembolization using DC Bead and doxorubicin hydrochloride. Chemoembolization repeats every 8 weeks for a total of 3 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline and at weeks 10 and 24.

Patients are followed at 4 weeks and then every 12 weeks thereafter.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 280 patients (140 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed hepatocellular carcinoma (HCC)

  * Advanced, unresectable disease
* No clinically significant ascites
* No modified Child-Pugh class C liver disease
* No main portal vein occlusion/involvement
* No extrahepatic tumor of any kind

PATIENT CHARACTERISTICS:

Age

* 18 and over (16 and over for patients residing in Scotland)

Performance status

* ECOG 0-2

Life expectancy

* More than 3 months

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Hemoglobin ≥ 8.5 g/dL
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin < 5.0 mg/dL
* Transaminases < 2.5 times upper limit of normal (ULN)
* INR < 1.5

Renal

* Creatinine < 2 times ULN

Cardiovascular

* No New York Heart Association class III or IV cardiac disease
* No acute angina
* No significant peripheral vascular disease
* No thrombosis of main portal vein
* LVEF ≥ 50%

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other concurrent serious medical condition
* No serious infection
* No psychological, familial, sociological, or geographical factors that would preclude study compliance
* No other malignancy within the past 5 years except carcinoma in situ of the cervix or non-melanoma skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior biologic therapy for advanced unresectable HCC

Chemotherapy

* No prior systemic or regional chemotherapy
* No prior chemotherapy for advanced unresectable HCC
* No other concurrent anticancer chemotherapy

Endocrine therapy

* No prior hormonal therapy for advanced unresectable HCC

Radiotherapy

* No prior radiotherapy for advanced unresectable HCC
* No other concurrent anticancer radiotherapy

Surgery

* More than 7 days since prior major surgery
* More than 3 days since prior laparoscopy

Other

* More than 4 weeks since prior investigational agents
* More than 6 weeks since prior ablative therapy and must have radiological evidence of progression if ablated site is the only site of disease
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2004-04

PRIMARY OUTCOMES:
Overall survival

SECONDARY OUTCOMES:
Overall response
Quality of life as assessed by EORTC QOL QLQ-30 and EORTC QLQ HCC18 at baseline and 10 and 24 weeks
Time to progression as assessed by RECIST criteria
Toxicity
Health economics
Proteomic and immunological analysis

CONTACTS AND LOCATIONS:
Overall Officials: O. J. Garden, Study Chair — Royal Infirmary of Edinburgh at Little France
Locations (10):
- United Kingdom (10):
  - Cancer Research UK Clinical Trials Unit - Birmingham, Birmingham, England
  - Bristol Haematology and Oncology Centre, Bristol, England
  - Addenbrooke's Hospital at Cambridge University Hospitals NHS Foundation Trust, Cambridge, England
  - Royal Liverpool University Hospital, Liverpool, England
  - Hammersmith Hospital, London, England
  - Freeman Hospital, Newcastle upon Tyne, England
  - Royal South Hants Hospital, Southampton, England
  - Royal Infirmary of Edinburgh at Little France, Edinburgh, Scotland
  - Royal Infirmary Edinburgh, Edinburgh, Scotland
  - West of Scotland Cancer Centre, Glasgow, Scotland